CLINICAL TRIAL: NCT02949115
Title: Acute and Chronic Effects of Red Beetroot Juice on High-Fat Meal-Induced Endothelial Dysfunction and Cardiometabolic Disturbances
Brief Title: Effects of Red Beetroot Juice on High-Fat Meal-Induced Endothelial Dysfunction and Cardiometabolic Disturbances
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Colorado State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sarah Johnson, Assistant Professor, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: COL00729
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Overweight; Obesity; Aging; Menopause
Keywords: Red beetroot; Dietary Nitrate; Polyphenols; Endothelial Function; High-Fat Meal; Overweight; Obesity; Aging; Cardiometabolic
MeSH Terms: conditions — Overweight; Obesity | interventions — Nitrates; potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 70 mL red beetroot juice (Experimental): 70 mL red beetroot juice naturally containing 300 mg nitrate.
  Interventions: Dietary Supplement: 70 mL red beetroot juice
- 70 mL placebo drink plus potassium nitrate (Active Comparator): 70 mL calorie-matched placebo control drink containing 489 mg potassium nitrate to deliver 300 mg nitrate.
  Interventions: Dietary Supplement: 70 mL placebo drink plus potassium nitrate
- 70 mL red beetroot juice without nitrate (Active Comparator): 70 mL red beetroot juice per day without nitrate.
  Interventions: Dietary Supplement: 70 mL red beetroot juice without nitrate
- 70 mL placebo drink (Placebo Comparator): 70 mL calorie-matched placebo control drink devoid of nitrate, vitamins, minerals, and polyphenols.
  Interventions: Dietary Supplement: 70 mL placebo drink

INTERVENTIONS:
Dietary Supplement: 70 mL red beetroot juice — 1x daily intake of 70 mL red beetroot juice
  Arms: 70 mL red beetroot juice
Dietary Supplement: 70 mL red beetroot juice without nitrate — 1x daily intake of 70 mL red beetroot juice without nitrate
  Arms: 70 mL red beetroot juice without nitrate
Dietary Supplement: 70 mL placebo drink plus potassium nitrate — 1x daily intake of 70 mL placebo control drink plus 489 mg potassium nitrate (300 mg nitrate)
  Arms: 70 mL placebo drink plus potassium nitrate
Dietary Supplement: 70 mL placebo drink — 1x daily intake of 70 mL placebo control drink
  Arms: 70 mL placebo drink

SUMMARY:
Aside from aging, numerous factors increase the risk for developing cardiovascular disease (CVD) including diet and nutrition. High-fat meal consumption induces postprandial vascular endothelial dysfunction and other cardiometabolic disturbances (e.g. dyslipidemia and hyperglycemia) in normal weight individuals and is exacerbated in overweight/obese individuals. These postprandial responses are likely largely due to activation of pro-inflammatory and pro-oxidant pathways. Given that much of the day is spent in the postprandial state, this may further impair cardiovascular health in aging overweight/obese individuals. Interventions that attenuate these responses are needed. Red beetroot (Beta vulgaris L.) is an excellent source of bioactive compounds including nitrate, flavonoids, phenolic acids, betalains, carotenoids, and ascorbic acid. These bioactive compounds and their metabolites have been shown to have antioxidative, anti-inflammatory, and cardiovascular-protective effects. These effects, particularly the cardiovascular-protective effects, have been primarily attributed to its high content of nitrate since it is converted to nitric oxide independent of the vascular endothelium via the enterosalivary nitrate-nitrite-nitric oxide pathway. However, red beetroot juice contains a number of other potentially beneficial bioactive compounds and few studies have aimed to determine whether these compounds work independently, additively, or synergistically in exerting these effects. Given the findings of previously conducted research in the broad area of red beetroot juice consumption and human health, it can be suggested that: 1) acute red beetroot juice consumption may prevent or attenuate the adverse postprandial responses to consuming a high-fat meal in individuals with exaggerated responses; and 2) chronic consumption of red beetroot may improve underlying factors contributing to these exaggerated responses. Accordingly, this project aims to: 1) investigate the efficacy of acute and chronic whole red beetroot juice consumption compared with its bioactive components in attenuating postprandial vascular endothelial dysfunction and adverse cardiometabolic responses to a high-fat meal; and 2) to gain insight into the underlying mechanisms responsible.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 4-period, 4-week crossover pilot clinical trial consisting of 2 postprandial tests for each period. Overweight or obese postmenopausal women and men aged 40 to 65 will be recruited from the greater Fort Collins, CO area. After telephone prescreening, participants will report to the study site for their first visit (Screening) where they will receive verbal and written explanation of the project, provide informed consent, followed by screening assessments. Qualified participants will be scheduled for a baseline visit and randomly assigned to their respective treatments. On the second visit (Baseline) following an overnight fast, anthropometrics and blood pressure will be measured and diet and physical activity records will be collected. Subjects will ingest their respective treatment 10 min prior to consuming the high-fat test meal. Various assessments will be performed and samples collected prior to and up to 4 hours post-meal consumption. At the third visit (Final), all assessments and sample collections will be repeated at the same time points but 24 hours after consuming the last dose of their respective treatments to test chronic rather than acute effects. Subjects will undergo a 4-week washout period before crossing over to the next treatment period. This will be repeated for all 4 treatments.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women and men
* BMI between 25 and 40 kg/m2

Exclusion Criteria:

* Hypertension, cardiovascular disease, diabetes, cancer, or kidney, liver, or pancreatic disease
* Individuals taking gastroesophageal reflux, antihypertensive, hypoglycemic, lipid-lowering, hormone replacement, erectile dysfunction medications or nitrates
* Participating in a weight loss program or actively trying to lose weight
* Smokers
* Heavy drinkers (> 3 drinks on any given occasion and/or > 7 drinks/week for women, or > 4 drinks on any given occasion and/or > 14 drinks/week for men)
* Allergy to meals/treatments
* Consuming > 2 servings red beetroot or beetroot juice/wk

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Vascular endothelial function | 0 and 4 hours post-meal consumption at baseline and 1 month for each treatment period.
  Vascular endothelial function will be assessed using reactive hyperemia index (EndoPAT) 0 and 4 hours post-meal consumption.

SECONDARY OUTCOMES:
Blood glucose, insulin, and indices of insulin sensitivity and resistance | 0 and 1, 2, and 4 hours post-meal consumption at baseline and 1 month for each treatment period.
  Blood glucose and insulin will be measured by biochemical analysis at 0 and 1, 2, and 4 hours post-meal consumption and indices of insulin sensitivity and resistance will be calculated.
Blood triglycerides | 0 and 1, 2, and 4 hours post-meal consumption at baseline and 1 month for each treatment period.
  Blood triglycerides will be measured by biochemical analysis at 0 and 1, 2, and 4 hours post-meal consumption.
Blood pressure | 0 and 1, 2, and 4 hours post-meal consumption at baseline and 1 month for each treatment period
  Peripheral and central blood pressure measured by an automatic sphygmomanometer and SphygmoCor at 0 and 1, 2, and 4 hours post-meal consumption.
Heart rate | 0 and 1, 2, and 4 hours post-meal consumption at baseline and 1 month for each treatment period.
  Heart rate will be measured by an automatic sphygmomanometer and SphygmoCor at 0 and 1, 2, and 4 hours post-meal consumption.
Arterial stiffness | Pre-meal consumption at baseline and 1 month for each treatment period.
  Arterial stiffness will be assessed as carotid-femoral pulse wave velocity and augmentation index (using SphygmCor and EndoPAT) at baseline and 1 month periods (pre-meal consumption).
Nitric oxide biomarkers | 0 and 1, 2, and 4 hours post-meal consumption at baseline and 1 month for each treatment period.
  Nitric oxide metabolites and molecules involved in nitric oxide production and bioavailability will be evaluated in saliva, blood, peripheral blood mononuclear cells, and biopsied venous endothelial cells at 0 and 1, 2, and 4 hours post-meal consumption.
Oxidative stress biomarkers | 0 and 4 hours post-meal consumption at baseline and 1 month for each treatment period.
  Biomarkers of oxidative stress will be evaluating in peripheral blood mononuclear cells and biopsied venous endothelial cells at 0 and 1, 2, and 4 hours post-meal consumption.
Pro-inflammatory biomarkers | 0 and 4 hours post-meal consumption at baseline and 1 month for each treatment period.
  Biomarkers of inflammation will be evaluating in peripheral blood mononuclear cells and biopsied venous endothelial cells at 0 and 4 hours post-meal consumption.

OTHER OUTCOMES:
Blood polyphenols and polyphenol metabolites | 0, 1, 2 and 4 hours post-meal consumption at baseline and 1 month for each treatment period.
  Blood polyphenols and metabolites will be measured by mass spectrometry at 0, 1, 2 and 4 hours post-meal consumption.
Urinary polyphenols and polyphenol metabolites | 0 and 24 hours post-meal consumption at baseline and 1 month for each treatment period.
  Urinary polyphenols and metabolites will be measured by mass spectrometry at 0 and 24 hours post-meal consumption.
Oral and gut microbiome | Pre-meal consumption at baseline and 1 month for each treatment period.
  The role of the oral and gut microbiome in efficacy of treatments at baseline and over time will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food Science and Human Nutrition, Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Litwin NS, Van Ark HJ, Hartley SC, Michell KA, Vazquez AR, Fischer EK, Melby CL, Weir TL, Wei Y, Rao S, Hildreth KL, Seals DR, Pagliassotti MJ, Johnson SA. Impact of Red Beetroot Juice on Vascular Endothelial Function and Cardiometabolic Responses to a High-Fat Meal in Middle-Aged/Older Adults with Overweight and Obesity: A Randomized, Double-Blind, Placebo-Controlled, Crossover Trial. Curr Dev Nutr. 2019 Oct 17;3(11):nzz113. doi: 10.1093/cdn/nzz113. eCollection 2019 Nov. PMID 31737860